CLINICAL TRIAL: NCT06920524
Title: Interest of a Musical Intervention on Stress Induced During Botulinum Toxin Injections in Spasticity
Brief Title: Interest of a Musical Intervention on Stress Induced During Botulinum Toxin Injections in Spasticity (MUSIBOT)
Acronym: MUSIBOT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RBHP 2024 BADIN; 2024-A02840-47 (Other: ANSM)
Record Dates: First submitted 2025-03-27; First posted 2025-04-09 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Stroke; Multiple Sclerosis; Spinal Cord Injury; Head Trauma Injury
Keywords: Musical intervention; Pain Management; stress; Botulinum toxin
MeSH Terms: conditions — Stroke; Multiple Sclerosis; Spinal Cord Injuries; Agnosia

STUDY DESIGN:
Intervention Model Description: At the first visit, consent will be obtained from the patient or guardian, followed by data collection (age, sex, pathology, date of first injection). Randomization will take place after this stage. All injections will follow the same protocol (tracking technique, MYOBOT 26G needle, ice analgesia on request). A Polar H10 heart rate monitor will measure the stress induced by the medical procedure. Before the injection, the patient will complete the STAI-Y1 anxiety questionnaire.The control group (CT-IM) will receive only the heart rate monitor, and will receive injections as usual. The intervention group (IM-IM) will be provided with a tablet and headphones to listen to selected music before the injection. At the end, all patients will rate their pain (VAS 0-10), anxiety (STAI-Y1) and satisfaction. Their perception of time will be compared with the actual duration of the medical procedure.At the second visit (M3±1 month), all patients will have access to music before the injection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group CT-IM : standard condition (No Intervention): The control group (CT-IM) will receive no special devices, apart from the Polar H10 heart rate monitor. This group will perform botulinum toxin injections as usual in the department, with the same assessments as the IM-IM group.
- Intervention group : IM-IM (Experimental): The intervention group (IM-IM) will receive a tablet and headphones to listen to music during the toxin injections. Then, during the waiting time, the patient, with or without assistance, will choose the music they wish to listen to, according to their musical tastes. The duration of the music can be modulated according to the duration of the medical procedure to follow.
  Interventions: Device: Intervention group IM-IM

INTERVENTIONS:
Device: Intervention group IM-IM — The intervention group (IM-IM) will receive a tablet and headphones to listen to music during the toxin injections. Then, during the waiting time, the patient, with or without assistance, will choose the music they wish to listen to, according to their musical tastes. The duration of the music can be modulated according to the duration of the medical procedure to follow.
  Arms: Intervention group : IM-IM

SUMMARY:
Botulinum toxin (BT) injections are a painful treatment frequently used to treat spasticity following central neurological damage (stroke, multiple sclerosis, spinal cord injury, head trauma). Tolerance of injections varies from patient to patient. For most patients, the pain experienced during the injection is a major source of stress.

Numerous clinical trials have demonstrated the role of music therapy in pain management. Music therapy uses a "U" shaped technique, allowing the patient to relax in different phases. This system has demonstrated beneficial effects on pain and anxiety in various fields, such as chronic and acute pain, Alzheimer's disease, fibromyalgia and neurological pain. Given the painful nature of spasticity and anxiety treatment, we aim to use a musical intervention to help patients cope better with injections.

The primary objective of the study is to investigate the effect of exposure to a musical intervention session during botulinum toxin injections, on injection-induced stress (heart rate variability).

Secondary objectives:

To study the effect of exposure to a musical intervention session during botulinum toxin injections, during the visit to injections #1, in terms of:

* Injection-induced stress for HRV parameters other than LF/HF
* Injection-induced pain
* Injection anxiety
* Patient satisfaction
* Effect of musical intervention on the medical procedure performed (botulinum toxin injections) expressed by the doctor at the end of the session.

To study the effect of exposure to a musical intervention session, during injections visit n°2, in order to evaluate the effect of repeated exposure to a musical intervention session, in terms of :

* Injection-induced stress for HRV parameters other than LF/HF
* Injection-induced pain
* Injection anxiety
* Patient satisfaction
* Effect of musical intervention on the medical procedure performed (botulinum toxin injections) expressed by the physician at the end of the session.

The hypothesis of this research is that a responsive musical intervention can, in adults, reduce the stress induced by botulinum toxin injections.

Patients will be selected from the cohort of patients regularly treated for botulinum toxin injections in the Physical and Rehabilitation Medicine (PRM) department at Clermont-Ferrand University Hospital. Botulinum toxin injections will take place in the PRM department. Each patient will participate in the study for a maximum of 4 months.

This study will be carried out in patients receiving regular botulinum toxin injections to treat spasticity. The first injection will be given with (IM-IM) or without musical intervention (CT-IM), depending on the randomization group, followed by the next injection with musical intervention. Patients will be able to choose the style of music (Jazz, Classical, Electronic, R&B, Ambient, Rock, etc.) that appeals to them in order to benefit from a minimum 20-minute session of musical intervention (duration varying according to the number of injections to be performed).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, male or female, suffering from spasticity of neurological origin (multiple sclerosis, stroke, head trauma, etc.) and eligible for botulinum toxin injection treatments.
* Patients with known pain and/or anxiety
* Able to give informed consent to participate in research
* Enrolled in a French Social Security system

Exclusion Criteria:

* Contraindication to musical intervention (severe hearing impairment, unstabilized psychotic disorders, history of auditory trauma)
* Major cognitive impairment
* Any medical condition deemed by the investigator to be incompatible with the research.
* Indication for MEOPA sedation during botulinum toxin injection sessions
* Medication or medical conditions likely to interfere with heart rate variability during the study: beta-blockers, anti-arrhythmics, anxiolytics, benzodiazepines, anti-hypertensives and calcium antagonists.
* Pregnant or breast-feeding women
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-04-25 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Stress | Baseline
  Patient stress, assessed during injection visit no. 1, estimated by the variation in heart rate variability (HRV), measured before and during the botulinum toxin injection session with the LF (sympathic activity)
Stress | Baseline
  Patient stress, assessed during injection visit no. 1, estimated by the variation in heart rate variability (HRV), measured before and during the botulinum toxin injection session with the HF parameter (parasympatic activity).
  The LF/HF ratio is a good reflection of the balance between sympathetic and parasympathetic nervous system activity, which can offer clues to stress regulation, cardiovascular health and physical adaptation. Thus, a low LF/HF ratio may be associated with better recovery, better emotional regulation, and a healthier balance of the autonomic nervous system.

SECONDARY OUTCOMES:
Stress | 3 months
  Patient stress during injection visit no. 2, estimated by the variation in heart rate variability (HRV), measured before and during the botulinum toxin injection session with the parameter LF/HF.
Intensity of pain | Baseline and 3 months
  The intensity of pain experienced by the patient during the botulinum toxin injection session, during visits to injections n°1 and n°2, measured by a simple numerical scale (ENS) ranging from 0 ("no pain") to 10 ("the worst pain imaginable") immediately after the end of the session.
Variation of anxiety | Baseline and 3 months
  Measurement of the variation in anxiety measured using the State Trait Anxiety Inventory-form Y Etat (STAI-Y1) self-questionnaire, during injection visits n°1 and n°2, before and after botulinum toxin injections. The STAI-Y1 questionnaire consists of 20 questions, measured on a Likert scale ranging from 1-" Not at all" to 4-"Very much so".
Measurement of perception of session time | Baseline and 3 months
  Measurement of perception of session time in relation to actual injection time at injection visits n°1 and n°2. Declarative data collected at the end of the session during the various visits.
Patient satisfaction with the procedure | Baseline and 3 months
  Patient satisfaction with the procedure assessed using a Visual Analogue Scale (VAS) ranging from 0 - "no satisfaction" to 10 - "highest satisfaction" measured after the injections, during injection visits n°1 and n°2.
Quality of the conditions under which botulinum toxin injections | Baseline and 3 months
  The quality of the conditions under which botulinum toxin injections were performed, as assessed by the doctor immediately after the end of the session for injections n°1 and n°2 [using a simple numerical scale (ENS) ranging from 0 ("extremely poor conditions") to 10 ("extremely good conditions")].

CONTACTS AND LOCATIONS:
Overall Officials: Marina BADIN, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Background] Guetin S, Portet F, Picot MC, Pommie C, Messaoudi M, Djabelkir L, Olsen AL, Cano MM, Lecourt E, Touchon J. Effect of music therapy on anxiety and depression in patients with Alzheimer's type dementia: randomised, controlled study. Dement Geriatr Cogn Disord. 2009;28(1):36-46. doi: 10.1159/000229024. Epub 2009 Jul 23. PMID 19628939
- [Background] Guétin S, Giniès P, Picot MC, et al. Évaluation et standardisation d'une nouvelle technique de musicothérapie dans la prise en charge de la douleur : le montage en " U ". Douleurs Eval - Diagn - Trait. 2010;11(5):213-218. doi:10.1016/j.douler.2010.06.001
- [Background] Guetin S, Brun L, Deniaud M, Clerc JM, Thayer JF, Koenig J. Smartphone-based Music Listening to Reduce Pain and Anxiety Before Coronarography: A Focus on Sex Differences. Altern Ther Health Med. 2016 Jul;22(4):60-3. PMID 27548494
- [Background] Bertacco M, Soyeux O, Durand R, Boudrias P, Wiseman L, Rompre P, Rainville P, Emami E, Gosselin N. Effect of personalized musical intervention on burden of care in dental implant surgery: A pilot randomized controlled trial. J Dent. 2022 May;120:104091. doi: 10.1016/j.jdent.2022.104091. Epub 2022 Mar 11. PMID 35283258
- [Background] Sorkpor SK, Montero-Hernandez S, Miao H, Pollonini L, Ahn H. Assessing the impact of preferred web app-based music-listening on pain processing at the central nervous level in older black adults with low back pain: An fNIRS study. Geriatr Nurs. 2023 Nov-Dec;54:135-143. doi: 10.1016/j.gerinurse.2023.09.005. Epub 2023 Oct 1. PMID 37782976
- [Background] Sorkpor SK, Miao H, Moore C, Johnson CM, Maria DMS, Pollonini L, Ahn H. Listening to Remotely Monitored Home-based Preferred Music for Pain in Older Black Adults with Low Back Pain: A Pilot Study of Feasibility and Acceptability. Pain Manag Nurs. 2023 Oct;24(5):e102-e108. doi: 10.1016/j.pmn.2023.07.001. Epub 2023 Jul 21. PMID 37482453
- [Derived] Angelvy P, Badin M, Pelletier-Visa M, Givron P, Pereira B, Coudeyre E. Musical intervention to reduce stress during botulinum toxin injection for spasticity: Protocol for a randomized controlled trial (MUSIBOT). PLoS One. 2025 Nov 25;20(11):e0327259. doi: 10.1371/journal.pone.0327259. eCollection 2025. PMID 41289288
- See also: Recommandations pour les médicaments. — https://ansm.sante.fr/documents/reference/recommandations-pour-les-medicaments